CLINICAL TRIAL: NCT04458896
Title: Stand When You Can: 6-week Pilot Study to Reduce Sedentary Time in Assisted Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lethbridge (Other)
Responsible Party: Principal Investigator, Dr. Jennifer Copeland, Professor, University of Lethbridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-001
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Sedentary Behavior; Aging
Keywords: assisted living; physical function; Social Ecological Model
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Non-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stand When You Can (Experimental): The intervention is grounded in Social Cognitive Theory and the Social Ecological Model (SEM). Multiple levels of the SEM will be targeted (individual, environmental, and organizational) over 6 weeks.
  Interventions: Behavioral: Stand When You Can

INTERVENTIONS:
Behavioral: Stand When You Can — Intervention strategies can be customized to different environments based on consultation with management. Some strategies will be mandatory:
  * Education session: group information session during the first week of the intervention (30min) to discuss sedentary time (ST), health risks, strategies to reduce ST, goal setting, & the identification of barriers and motivators to reducing ST. Group discussion will be encouraged to increase self-motivation and self-efficacy. An information "workbook" will be given to each attendee for their personal use and goal setting.
  * Point of decision prompts (ie: signs that encourage standing; see attachments) will be placed in common areas of the facility, and/or given as pamphlets to residents.
  * An intervention package will be provided to the Activity Coordinator and Manager of the facility. This package will provide an introductory letter along with materials to promote reduced sedentary time in the facility

SUMMARY:
Prolonged daily sedentary time is associated with increased risk of cardiometabolic diseases, impaired physical function, and mortality. Older adults are more sedentary than any other age group and those in assisted living residences accumulate even more sedentary time as they often have little need to engage in light-intensity or standing activities such as cleaning or meal preparation. This "low movement" environment can hasten functional decline. Thus, the purpose of this study was to develop a multi-level intervention to reduce and interrupt sedentary time within assisted living residences and conduct a pilot study to determine if the intervention is feasible and if further testing is warranted.

DETAILED DESCRIPTION:
This is a voluntary single-arm uncontrolled trial in assisted living residences. Pre- and post- intervention assessments will be conducted over two sessions; the intervention period is 6 weeks.

First session:

In the first session participants will complete informed consent, compete all questionnaires, and be fitted with the active PALs for measuring sedentary time. This should take approximately 30-60 minutes. The second session will be 7 days later, and the investigators will retrieve the ActivPAL inclinometer and then complete the Short Performance Physical Battery. This should take 20-30 minutes. Health-related quality of Life will be assessed using the Euro Quality of Life 5 dimension questionnaire (EQ-5D). This is a generic health status questionnaire (i.e. it is not disease specific) and consists of a descriptive system and a visual analogue scale (VAS). Five dimensions are included: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It is widely used and has good reliability. General Quality of Life will be assessed using the ICEpop CAPability measure for Older people (ICECAP-O). The ICECAP-O has a broad view of quality of life and covers the domains of attachment (love and friendship), security (thinking about the future without concern), role (doing things that make participants feel valued), enjoyment (enjoyment and pleasure), and control (independence). Both questionnaires are attached and the estimated time for completion is about 10 minutes.Sedentary time will be with an activPAL4™ inclinometer and the Longitudinal Aging Study Amsterdam (LASA) self-report sedentary behaviour questionnaire. The activPAL4™ device is enclosed in a nitrile sleeve and secured to the thigh using medical tape. Skin will be monitored for irritation. Both the finger cots and the nitrile sleeves are single use. The activPAL4™ inclinometers are only 9 grams and 5mm thick, making them comfortable for 7-day wear on the thigh. Using proprietary algorithms and software, it classifies an individual's free-living activity into periods spent sleeping, sitting, standing and ambulating as well as step counts, activity start time and activity duration. This allows for quantification of these movement behaviours over 24 hours. The unit will be worn for 7 days to determine the pre-intervention movement profile. Mid-way through the 7 day period researchers will check in with participants to ensure there are no problems. These devices have been used extensively with older adults in previous research.

The LASA sedentary behavior questionnaire is moderately associated with accelerometer-measured sedentary time (r=.46) and reliably ranks sedentary time in older adults. While self-report tools underestimate total sedentary time, they provide valuable information about the context (eg. where or with whom) and type (eg. reading or watching TV) of sedentary behaviours, which will be valuable for evaluating the intervention. (See attachments for a copy of the questionnaire).

Second Session:

Blood pressure in mmHg and heart rate in beats per minute will be measured at rest in a seated position. If Blood Pressure exceeds 160/90 mmHg or heart rate exceeds 99 beats per minute, the participants will not complete the SPPB described below. These will be measured using an automated sphygmomanometer. Height in centimetres and weight in kilograms will be measured using an electronic scale and stadiometer.Participants will be asked to refrain from smoking or consuming caffeine for 2 hours before the appointment and avoid exercise or strenuous physical activity the day of the assessment. The Short Performance Physical Battery (SPPB) will be used to assess physical function. The SPPB is an objective assessment tool for evaluating lower extremity functioning in older persons and it includes assessments of gait speed, standing balance, and timed chair rises (see attachment for details). It was developed by the National Institute on Aging and has been shown to have high validity and reliability in measuring physical function in older adults. The participants will also measure grip strength by having participants grasp a hand grip dynamometer and squeezing as hard as possible, with each hand. The entire battery of tests will be conducted in a circuit format and will take ≤20 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* independently mobile residents of assisted living communities 65 years or older
* able to read and write in English
* able to provide informed consent

Exclusion Criteria:

* do not have a diagnosed cognitive impairment
* expecting to have a medical procedure that would require more than 1 week of rest during the intervention period

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Daily time spent sedentary measured by activPAL4™ inclinometers | 6 weeks
  Sedentary time in minutes per day will be assessed with the activPAL4™ inclinometer which measures movement patterns and body posture 24 hours/day and can monitor body positions, making them useful for measuring sedentary time. activPALs have been found to be valid and reliable in comparison to direct observation (R2 = 0.94). The activPAL4s were waterproofed using a nitrile sleeve and affixed to the thigh using Tegaderm (3M Medical, USA).
Physical function of The lower extremities measured by the Short Physical Performance Battery | 6 weeks
  The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older adults and it includes assessments of gait speed (4 m walk), standing balance (side by side, semi-tandem, and tandem), and 5 timed chair rises. The SPPB has been shown to have good predictive and concurrent validity and reliability (intraclass correlation coefficient > 0.70) in measuring physical function in older adults and is also predictive of mobility impairment. A maximum score of 12 represents good physical function.
Quality of Life measured by the EQ-5D-5L | 6 weeks
  The EQ-5D-5L is a generic measure of health status that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, along a five-point scale (no problems, slight problems, moderate, severe, and unable to do the action/extreme). These questions create a health state which will be translated to a summary index value using the Crosswalk Index Value Calculator (US values, euroqol.org). A value of 1 represents the best possible health state, with health states diminishing as they approach zero. It also includes a visual analogue scale for overall health anchored between 0 (worst health imaginable) to 100 (best health imaginable). The EQ-5D-5L has a discriminatory power of 0.68 and a test-retest reliability of 0.69.
Upper body strength measured by grip strength | 6 weeks
  Grip strength will be measured in kilograms using a dynamometer (Creative Health Products Inc, USA) following Canadian Society of Exercise Physiology testing guidelines. Two trials will be completed by either hand and the best score from either hand will be combined into one score. A higher score represents better strength.
Quality of Life measured by the ICEpop CAPability Measure for Older People Scale | 6 weeks
  The ICECAP-O is a broader measure of quality of life that does not focus on physical health but covers the domains of attachment, security, role, enjoyment, and control. The ICECAP-O has been shown to be reliable and have good construct validity as a measure of quality of life. A score is calculated between 0 and 1 with 0 representing no capability (e.g. death) and 1 representing maximum capability.
Self-reported time spent in sedentary behaviour measured by the LASA Sedentary Behaviour Questionnaire | 6 weeks
  The Longitudinal Aging Study Amsterdam (LASA) Sedentary Behaviour Questionnaire estimates self-reported sedentary time by asking participants about time (hours:minutes) spent in 10 sitting behaviours on an average weekday or weekend day. The questionnaire has a test-retest reliability of 0.71 (95% CI 0.57-0.81) but may underestimate total sedentary time by as much as 2.1 hours. The six domains of napping, reading, listening to music, watching TV, engaging in seated hobbies, and talking to friends had the highest correlation with device-measured sedentary time. Thus, the investigators will only include these six domains when calculating self-reported sedentary time.

SECONDARY OUTCOMES:
Program feasibility | 6 weeks
  The investigators will collect feedback forms from residents after the 6-week intervention to gain an understanding of which strategies were used most frequently and how much they liked or disliked the different components of the intervention. Survey responses will be displayed in frequency tables.
Program Feedback Interviews with Staff | 6 weeks
  The investigators will interview the staff to receive staff feedback about ways the program could improve for future iterations. Feedback questions include what components seem to resonate with residents, which components were not utilized, and any other strategies the investigators could leverage to improve delivery and support. All staff will provide written informed consent prior to the interview.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Copeland, PhD, Principal Investigator — University of Lethbridge
Locations (1):
- University of Lethbridge, Lethbridge, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data of device-measured and self-reported sedentary time, physical function and quality of life measures
Time Frame: 10 years (2030)
Access Criteria: Email Dr. Copeland for access

REFERENCES:
- [Derived] Voss ML, Pope JP, Larouche R, Copeland JL. Stand When You Can: development and pilot testing of an intervention to reduce sedentary time in assisted living. BMC Geriatr. 2020 Aug 6;20(1):277. doi: 10.1186/s12877-020-01647-z. PMID 32762644